CLINICAL TRIAL: NCT02534896
Title: To Evaluate The Efficacy And Safety Of Sunpharma1505 Compared With Reference1505 In Subjects With Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLR_15_05
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Active Rheumatoid Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment 1: Sunpharma1505 (Low dose) and Placebo (Experimental)
  Interventions: Drug: Treatment I
- Treatment II: Sunpharma1505 (High Dose) and Placebo (Experimental)
  Interventions: Drug: Treatment II
- Treatment III: Reference1505 and Placebo (Active Comparator)
  Interventions: Drug: Treatment III

INTERVENTIONS:
Drug: Treatment I — Sunpharma1505 and Placebo
  Arms: Treatment 1: Sunpharma1505 (Low dose) and Placebo
Drug: Treatment II — Sunpharma1505 and Placebo
  Arms: Treatment II: Sunpharma1505 (High Dose) and Placebo
Drug: Treatment III — Reference1505 and Placebo
  Arms: Treatment III: Reference1505 and Placebo

SUMMARY:
This study is designated to evaluate the safety and efficacy of Sunpharma1505 in subjects with active rheumatoid arthritis who are experiencing a flare/exacerbation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able and willing to give written informed consent and is available for entire study.
2. Male or female ≥ 18 years old
3. Willing and able to comply with the study protocol visits, assessments and accessible for follow up
4. Known Diagnosed Rheumatoid arthritis
5. Subjects of child bearing potential should be non-lactating and must be practicing an acceptable method of birth control as judged by the Investigator

Exclusion Criteria:

1. Subjects who are pregnant or intend to become pregnant during the study
2. Subject with positive hepatitis panel and / or anti-hepatitis B core antibodies, and / or hepatitis C virus antibody [anti-HCV]), and / or a positive Human immunodeficiency virus (HIV) antibody.
3. Known sensitivity to any component of the study drug or previous hypersensitivity reaction or other clinically significant reaction to IV medications, biologic therapy or IV radiocontrast agents.
4. Active infection requiring systemic treatment
5. Planned surgery during the study period or had undergone major surgery within the 60 Days prior to the Screening visit.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-11; Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- Belgium (8):
  - Sun Pharma Site 17, Brussels
  - Sun Pharma Site 18, Brussels
  - Sun Pharma Site 21, Brussels
  - Sun Pharma Site 22, Brussels
  - Sun Pharma Site 23, Brussels
  - Sun Pharma Site 16, Leuven
  - Sun Pharma Site 19, Liège
  - Sun Pharma Site 20, Merksem
- Netherlands (12):
  - Sun Pharma Site 11, Amsterdam
  - Sun Pharma Site 9, Amsterdam
  - Sun Pharma Site 6, Enschede
  - Sun Pharma Site 4, Heerlen
  - Sun Pharma Site 7, Hilversum
  - Sun Pharma Site 2, Leeuwarden
  - Sun Pharma Site 8, Lelystad
  - Sun Pharma Site 10, Rotterdam
  - Sun Pharma Site 3, Rotterdam
  - Sun Pharma Site 5, Sneek
  - Sun Pharma Site 14, Uden
  - Sun pharma Site 01, Utrecht

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment I : Sunpharma1505 (Low Dose) and Placebo; Treatment II: Sunpharma1505 (High Dose) and Placebo; Treatment III: Reference1505 and Placebo: solution for injection/infusion Day 1 and 15
Period: Overall Study
Arm/Group | Treatment I : Sunpharma1505 (Low Dose) and Placebo | Treatment II: Sunpharma1505 (High Dose) and Placebo | Treatment III: Reference1505 and Placebo
Started | 49 | 52 | 49
Completed | 45 | 51 | 48
Not Completed | 4 | 1 | 1
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Insufficient therapeutic response | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment I: Sunpharma1505 (Low Dose) and Placebo; Treatment II: Sunpharma1505 (High Dose) and Placebo; Treatment III: Reference1505 and Placebo: solution for injection/infusion Day 1 and 15
- Total: Total of all reporting groups
Arm/Group | Treatment I: Sunpharma1505 (Low Dose) and Placebo | Treatment II: Sunpharma1505 (High Dose) and Placebo | Treatment III: Reference1505 and Placebo | Total
Number analyzed (Participants) | 49 | 52 | 49 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (13.79) | 56.4 (10.74) | 56.7 (11.18) | 56.1 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 42 | 35 | 115
  Male | 11 | 10 | 14 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 46 | 49 | 43 | 138
  More than one race | 1 | 1 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Good/Moderate European League Against Rheumatism Responders
Time Frame: week 1
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment I : Sunpharma1505 (Low Dose) and Placebo | Treatment II: Sunpharma1505 (High Dose) and Placebo | Treatment III: Reference1505 and Placebo
Number analyzed (Participants) | 49 | 52 | 49
Participants | 42 | 45 | 32
Statistical Analysis 1: Comparison: Treatment I : Sunpharma1505 (Low Dose) and Placebo vs Treatment III: Reference1505 and Placebo; Test type: Superiority; p = 0.018, Hochberg and Gatekeeping
Statistical Analysis 2: Comparison: Treatment II: Sunpharma1505 (High Dose) and Placebo vs Treatment III: Reference1505 and Placebo; Test type: Superiority; p = 0.007, Hochberg and Gatekeeping

2. Secondary Outcome: Good European League Against Rheumatism -Responders
Time Frame: Day 8
Population: intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment I : Sunpharma1505 (Low Dose) and Placebo | Treatment II: Sunpharma1505 (High Dose) and Placebo | Treatment III: Reference1505 and Placebo
Number analyzed (Participants) | 49 | 52 | 49
Participants | 21 | 26 | 10
Statistical Analysis 1: Comparison: Treatment I : Sunpharma1505 (Low Dose) and Placebo vs Treatment III: Reference1505 and Placebo; Test type: Superiority; p = 0.028, Hochberg and Gatekeeping
Statistical Analysis 2: Comparison: Treatment II: Sunpharma1505 (High Dose) and Placebo vs Treatment III: Reference1505 and Placebo; Test type: Superiority; p = 0.003, Hochberg and Gatekeeping

3. Secondary Outcome: Good/Moderate European League Against Rheumatism Responders
Time Frame: Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment I : Sunpharma1505 (Low Dose) and Placebo | Treatment II: Sunpharma1505 (High Dose) and Placebo | Treatment III: Reference1505 and Placebo
Number analyzed (Participants) | 49 | 52 | 49
Participants | 42 | 43 | 42
Statistical Analysis 1: Comparison: Treatment I : Sunpharma1505 (Low Dose) and Placebo vs Treatment III: Reference1505 and Placebo; Test type: Superiority; p = 0.960, Hochberg and Gatekeeping
Statistical Analysis 2: Comparison: Treatment II: Sunpharma1505 (High Dose) and Placebo vs Treatment III: Reference1505 and Placebo; Test type: Superiority; p = 0.339, Hochberg and Gatekeeping

4. Secondary Outcome: Good European League Against Rheumatism Responders
Time Frame: Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment I : Sunpharma1505 (Low Dose) and Placebo | Treatment II: Sunpharma1505 (High Dose) and Placebo | Treatment III: Reference1505 and Placebo
Number analyzed (Participants) | 49 | 52 | 49
Participants | 24 | 33 | 21
Statistical Analysis 1: Comparison: Treatment I : Sunpharma1505 (Low Dose) and Placebo vs Treatment III: Reference1505 and Placebo; Test type: Superiority; p = 0.573, Hochberg and Gatekeeping
Statistical Analysis 2: Comparison: Treatment II: Sunpharma1505 (High Dose) and Placebo vs Treatment III: Reference1505 and Placebo; Test type: Superiority; p = 0.374, Hochberg and Gatekeeping

ADVERSE EVENTS:
Time Frame: Week 12
Groups:
- Treatment I: Sunpharma1505 (Low Dose) and Placebo: Treatment I: Treatment I and Placebo
- Treatment II: Sunpharma1505 (High Dose) and Placebo: Treatment II: Treatment II and Placebo
- Treatment III: Reference1505 and Placebo: Treatment III: Treatment III and Placebo
Arm/Group | Treatment I: Sunpharma1505 (Low Dose) and Placebo | Treatment II: Sunpharma1505 (High Dose) and Placebo | Treatment III: Reference1505 and Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 4/49 | 1/52 | 2/49
Other Adverse Events (participants affected / at risk) | 42/49 | 46/52 | 39/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment I: Sunpharma1505 (Low Dose) and Placebo (N=49) | Treatment II: Sunpharma1505 (High Dose) and Placebo (N=52) | Treatment III: Reference1505 and Placebo (N=49)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment I: Sunpharma1505 (Low Dose) and Placebo (N=49) | Treatment II: Sunpharma1505 (High Dose) and Placebo (N=52) | Treatment III: Reference1505 and Placebo (N=49)
Hot flush (Vascular disorders) | 4 | 6 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4
Dizziness (Nervous system disorders) | 4 | 2 | 2
Fatigue (General disorders) | 6 | 6 | 5
Nausea (Gastrointestinal disorders) | 9 | 6 | 1
Nasopharyngitis (Infections and infestations) | 6 | 5 | 4
Headache (Nervous system disorders) | 8 | 9 | 6
Influenza (Infections and infestations) | 3 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4
Hyeprhidrosis (Skin and subcutaneous tissue disorders) | 1 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT02534896/Prot_SAP_000.pdf